CLINICAL TRIAL: NCT01492218
Title: A Prospective, Open-labelled, Non-controlled Observational Study to Assess Patient Satisfaction, Physician Acceptability and Safety of Mixtard® 30 NovoLet® for the Treatment of Diabetes Mellitus
Brief Title: Observational Study With Mixtard® 30 NovoLet® to Assess Patient Satisfaction
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-1885
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — biphasic human insulin 30

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoLet®
  Interventions: Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic human insulin 30 — Administered via the NovoLet® device and according to the instructions in the product insert or as instructed by the physician. Individually adjusted dosage as instructed by the physician.

SUMMARY:
This study is conducted in Asia. The aim of this study is to assess patient satisfaction after switching to biphasic human insulin 30 treatment using the NovoLet® insulin device as treatment for diabetes mellitus under normal clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or type 2)
* Patient not presently using Mixtard® 30 NovoLet®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with type 1 or type 2 diabetes mellitus and are not presently using Mixtard® 30 NovoLet®
Sampling Method: Probability Sample
Enrollment: 1330 (Actual)
Dates: Start 2004-03-15 (Actual); Primary Completion 2004-08-30 (Actual); Study Completion 2004-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) score

SECONDARY OUTCOMES:
Adverse events
Technical complaints of NovoLet® device

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manila, Philippines

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com